CLINICAL TRIAL: NCT07353658
Title: The Effect of Intermittent Versus Continuous Enteral Feeding on Outcomes in Severe Stroke: An Exploratory Study
Brief Title: Effect of Intermittent Enteral Feeding in Severe Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20252538jiangwen
Record Dates: First submitted 2025-12-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Severe Stroke; Enteral Nutrition
Keywords: Stroke; Enteral Nutrition
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Enteral Nutrition Group (Experimental)
  Interventions: Behavioral: Intermittent Enteral Feeding
- Continuous Enteral Nutrition Group (Active Comparator)
  Interventions: Behavioral: Continuous Enteral Feeding

INTERVENTIONS:
Behavioral: Intermittent Enteral Feeding — Participants randomized to this group will receive enteral nutrition via a nasogastric or nasojejunal tube using an intermittent, daytime-only feeding schedule designed to align with the physiological circadian rhythm.
  Arms: Intermittent Enteral Nutrition Group
Behavioral: Continuous Enteral Feeding — Participants randomized to this group will receive enteral nutrition via a nasogastric or nasojejunal tube using the standard, continuous 24-hour feeding method commonly employed in critical care settings.
  Arms: Continuous Enteral Nutrition Group

SUMMARY:
This is a single-center, randomized, exploratory clinical trial investigating whether intermittent enteral feeding improves outcomes compared to continuous feeding in patients with severe stroke. The study will enroll 60 patients to evaluate the impact on 90-day all-cause mortality, neurological function, nutritional status, and safety. It will also explore underlying mechanisms through analysis of metabolic profiles, circadian gene expression, and gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. It was definitely diagnosed as acute stroke by clinical imaging.
3. Enteral nutrition program can be started within 72 hours of onset.
4. Baseline GCS≤12 or NIHSS≥11
5. There is nutritional risk (NRS 2002≥3), Wadian drinking water test≥ 3 or there is consciousnessdisorder,it is estimated that you need to receive nutritional support treatment for ≥7 days
6. Obtain informed consent

Exclusion Criteria:

1. Before joining the group, he had received total parenteral nutrition treatment.
2. There are contraindications to enteral nutrition.
3. Unstable vital signs
4. Dementia or severe disability before onset (mRS≥3)
5. There are concomitant diseases that will interfere with outcome evaluation and/or follow-up.
6. Participating in other interventional clinical trials.
7. Other circumstances in which the study cannot be completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 90 days post-randomization

SECONDARY OUTCOMES:
90-day unfavorable outcome rate | at 90 days
  Defined as a modified Rankin Scale (mRS) score of 3-6
Neurological deficit score | at Day 3 and Day 7 post-randomization
  National Institutes of Health Stroke Scale (NIHSS) score
Activities of daily living | 90 days post-randomization
  Barthel Index (BI)
Nutritional status indicators | Baseline and Day 7 assessments
  Serum albumin (ALB); Serum prealbumin (PAB); Serum total protein (TP); Hemoglobin (HB) levels; Mid-upper arm circumference (MUAC); Triceps skinfold thickness (TSF)
Incidence of gastrointestinal intolerance | Throughout the intervention period (expected ≥7 days)
  Gastric retention; diarrhea; constipation and gastrointestinal bleeding
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Throughout the study period (up to 90-day follow-up).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reignier J, Plantefeve G, Mira JP, Argaud L, Asfar P, Aissaoui N, Badie J, Botoc NV, Brisard L, Bui HN, Chatellier D, Chauvelot L, Combes A, Cracco C, Darmon M, Das V, Debarre M, Delbove A, Devaquet J, Dumont LM, Gontier O, Groyer S, Guerin L, Guidet B, Hourmant Y, Jaber S, Lambiotte F, Leroy C, Letocart P, Madeux B, Maizel J, Martinet O, Martino F, Maxime V, Mercier E, Nay MA, Nseir S, Oziel J, Picard W, Piton G, Quenot JP, Reizine F, Renault A, Richecoeur J, Rigaud JP, Schneider F, Silva D, Sirodot M, Souweine B, Tamion F, Terzi N, Thevenin D, Thiery G, Thieulot-Rolin N, Timsit JF, Tinturier F, Tirot P, Vanderlinden T, Vinatier I, Vinsonneau C, Voicu S, Lascarrou JB, Le Gouge A; NUTRIREA-3 Trial Investigators; Clinical Research in Intensive Care; Sepsis (CRICS-TRIGGERSEP)Group. Low versus standard calorie and protein feeding in ventilated adults with shock: a randomised, controlled, multicentre, open-label, parallel-group trial (NUTRIREA-3). Lancet Respir Med. 2023 Jul;11(7):602-612. doi: 10.1016/S2213-2600(23)00092-9. Epub 2023 Mar 20. PMID 36958363
- [Result] Zhao J, Yuan F, Song C, Yin R, Chang M, Zhang W, Zhang B, Yu L, Jia Y, Ma Y, Song Y, Wang C, Song C, Wang X, Shang L, Yang F, Jiang W; OPENS Trial Investigators. Safety and efficacy of three enteral feeding strategies in patients with severe stroke in China (OPENS): a multicentre, prospective, randomised, open-label, blinded-endpoint trial. Lancet Neurol. 2022 Apr;21(4):319-328. doi: 10.1016/S1474-4422(22)00010-2. Epub 2022 Feb 24. PMID 35219379
- [Result] Panwar R, Kumar N, Parikh H, Dash S, Rai S. Standard continuous feeding versus intermittent feeding among mechanically ventilated patients in intensive care: A systematic review and meta-analysis of randomized controlled trials. Clin Nutr. 2025 Aug;51:40-49. doi: 10.1016/j.clnu.2025.05.024. Epub 2025 Jun 7. PMID 40516326
- [Result] Zhu W, Jiang Y, Li J. Intermittent versus continuous tube feeding in patients with hemorrhagic stroke: a randomized controlled clinical trial. Eur J Clin Nutr. 2020 Oct;74(10):1420-1427. doi: 10.1038/s41430-020-0579-6. Epub 2020 Mar 9. PMID 32152512
- [Result] Arabi YM, Aldawood AS, Haddad SH, Al-Dorzi HM, Tamim HM, Jones G, Mehta S, McIntyre L, Solaiman O, Sakkijha MH, Sadat M, Afesh L; PermiT Trial Group. Permissive Underfeeding or Standard Enteral Feeding in Critically Ill Adults. N Engl J Med. 2015 Jun 18;372(25):2398-408. doi: 10.1056/NEJMoa1502826. Epub 2015 May 20. Erratum In: N Engl J Med. 2015 Sep 24;373(13):1281. doi: 10.1056/NEJMx150028. PMID 25992505
- [Result] Heyland DK, Cahill N, Day AG. Optimal amount of calories for critically ill patients: depends on how you slice the cake! Crit Care Med. 2011 Dec;39(12):2619-26. doi: 10.1097/CCM.0b013e318226641d. PMID 21705881
- [Result] Wong HJ, Harith S, Lua PL, Ibrahim KA. Prevalence and Predictors of Malnutrition Risk among Post-Stroke Patients in Outpatient Setting: A Cross-Sectional Study. Malays J Med Sci. 2020 Jul;27(4):72-84. doi: 10.21315/mjms2020.27.4.7. Epub 2020 Aug 19. PMID 32863747
- [Result] van Wijk N, Studer B, van den Berg CA, Ripken D, Lansink M, Siebler M, Schmidt-Wilcke T. Evident lower blood levels of multiple nutritional compounds and highly prevalent malnutrition in sub-acute stroke patients with or without dysphagia. Front Neurol. 2023 Jan 10;13:1028991. doi: 10.3389/fneur.2022.1028991. eCollection 2022. PMID 36703642
- [Result] Sharie SA, Almari R, Azzam S, Al-Husinat L, Araydah M, Battaglini D, Schultz MJ, Patroniti NA, Rocco PR, Robba C. Brain Protective Ventilation Strategies in Severe Acute Brain Injury. Curr Neurol Neurosci Rep. 2025 Oct 13;25(1):68. doi: 10.1007/s11910-025-01462-2. PMID 41082009
- [Result] Ma Q, Li R, Wang L, Yin P, Wang Y, Yan C, Ren Y, Qian Z, Vaughn MG, McMillin SE, Hay SI, Naghavi M, Cai M, Wang C, Zhang Z, Zhou M, Lin H, Yang Y. Temporal trend and attributable risk factors of stroke burden in China, 1990-2019: an analysis for the Global Burden of Disease Study 2019. Lancet Public Health. 2021 Dec;6(12):e897-e906. doi: 10.1016/S2468-2667(21)00228-0. PMID 34838196
- [Result] GBD 2021 Stroke Risk Factor Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2021: a systematic analysis for the Global Burden of Disease Study 2021. Lancet Neurol. 2024 Oct;23(10):973-1003. doi: 10.1016/S1474-4422(24)00369-7. PMID 39304265
- [Result] Walter K. What Is Acute Ischemic Stroke? JAMA. 2022 Mar 1;327(9):885. doi: 10.1001/jama.2022.1420. No abstract available. PMID 35230392